CLINICAL TRIAL: NCT02514434
Title: Usefulness of Non-contrast MagnetIc Resonance imAging Versus Non-Contrast Ultrasonography for surveiLlancE of HepatoCellular Carcinoma [MIRACLE-HCC]
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 4-2015-0029
Record Dates: First submitted 2015-07-23; First posted 2015-08-03 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Compensated Liver Cirrhosis
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasonography (Experimental): Subjects will be regularly screened for HCC by ultrasonography with serum AFP(alpha fetoprotein).
  Interventions: Radiation: Ultrasonography
- Non-contrast MRI (Experimental): Subjects will be regularly screened for HCC by non-contrast magnetic resonance imaging(MRI) with serum AFP(alpha fetoprotein).
  Interventions: Radiation: non-contrast MRI

INTERVENTIONS:
Radiation: Ultrasonography — Subjects will be randomly allocated to either Ultrasonography arm or Non-contrast MRI arm for their surveillance method.
  Arms: Ultrasonography
Radiation: non-contrast MRI — Subjects will be randomly allocated to either Ultrasonography arm or Non-contrast MRI arm for their surveillance method.
  Arms: Non-contrast MRI

SUMMARY:
The investigators will investigate the usefulness of ultrasonography versus non-contrast magnetic resonance imaging for surveillance of hepatocellular carcinoma through this prospective, randomized trial.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the major complications in patients with chronic liver disease. The prognosis of HCC relies on the extent of disease at the time of diagnosis. Hence to detect cancer at an earlier stage, a regular surveillance test is important for the subjects with a high risk of developing cancer. Current guidelines recommend a regular surveillance using ultrasonography at a 6 month-interval. Ultrasonography is a non-invasive and safe procedure, yet it is limited by the skills of the operator and it is often difficult to differentiate cancer from regenerating nodules especially in atrophied cirrhotic liver. According to a recent meta-analysis, the overall sensitivity and specificity of detecting liver cancer using ultrasonography were both over 90%, however the sensitivity was decreased to 60% in detecting early lesions in which surgery or liver transplantation is indicated. Of note, addition of AFP to ultrasonography also failed to increase the sensitivity in detecting small cancers. Taken together, there is a need to develop a new surveillance test with an improved sensitivity and specificity.

Recently, a retrospective study reported that CT or MRI showed a better sensitivity than ultrasonography in detecting early liver cancer. However, performing CT as a surveillance test is limited by frequent exposure to radiation and contrast-dye agent. Although MRI does not have the risk of radiation-exposure, it is limited by the high cost. On the contrast, non-contrast MRI offers a cost that is comparable to US and an absence of exposure to radiation or contrast-dye agent, which suggests non-contrast MRI as a good alternative surveillance tool for early detection of HCC. Therefore, in this prospective, randomized trial, the investigators will investigate the usefulness of ultrasonography versus non-contrast magnetic resonance imaging for surveillance of hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject between 20 and 70 years of age at the time of randomization
* Has chronic liver disease with compensated liver cirrhosis (Child-Pugh score A), defined as 1) histologically confirmed cirrhosis, or 2) has chronic liver disease and shows the presence of splenomegaly or other typical findings of liver cirrhosis on ultrasonography, computed tomography, or magnetic resonance imaging, or 3) has chronic liver disease and shows the presence of endoscopically-confirmed esophageal or gastric varices
* Absence of severe cardiovascular, pulmonary, renal or infectious diseases, other than chronic liver disease
* Absence of a history of malignancy within previous 5 years
* Can and will comply with the requirements of the protocol (e.g. return for follow-up visits), in the opinion of the investigator
* Has provided written informed consent

Exclusion Criteria:

* Greater than 70 years of age
* Presence of liver cancer or other intrahepatic malignancy
* Has a history of malignancy within previous 5 years
* Is pregnant or breast-feeding

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2015-03-30 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Tumor stage of HCC | 6 months
  Comparing tumor stage and resectability rate of HCC between participants undergoing HCC surveillance using ultrasonography and non-contrast MRI.
Resectability rate of HCC | 6 months
  Comparing tumor stage and resectability rate of HCC between participants undergoing HCC surveillance using ultrasonography and non-contrast MRI.

SECONDARY OUTCOMES:
Five-year overall survival | 5 years after the study enrollment
Liver-related mortality | 5 years after the study enrollment
Post-treatment recurrence rate | 5 years after the study enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Gastroenterology, Department of Internal Medicine, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Rhee H, Kim MJ, Kim DY, An C, Kang W, Han K, Roh YH, Han KH, Ahn SH, Choi JY, Park JY, Chung YE, Kim SU, Kim BK, Lee S, Lee HW, Lee JS. Noncontrast Magnetic Resonance Imaging vs Ultrasonography for Hepatocellular Carcinoma Surveillance: A Randomized, Single-Center Trial. Gastroenterology. 2025 Jun;168(6):1170-1177.e12. doi: 10.1053/j.gastro.2024.12.035. Epub 2025 Jan 22. PMID 39855314
- [Derived] An C, Kim DY, Choi JY, Han KH, Roh YH, Kim MJ. Noncontrast magnetic resonance imaging versus ultrasonography for hepatocellular carcinoma surveillance (MIRACLE-HCC): study protocol for a prospective randomized trial. BMC Cancer. 2018 Sep 24;18(1):915. doi: 10.1186/s12885-018-4827-2. PMID 30249190